CLINICAL TRIAL: NCT07184216
Title: Effect of a Person-Centred Care Intervention for Families Providing Home-Based Care to a Person With Advanced Chronic Illness: A Pilot Randomised Controlled Trial
Acronym: HELP-F
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: University of Navarra (Other); Navarre Health Research Institute (IdiSNA), Spain (Unknown); University of Gothenburg Center for Person-Centred Care, GPCC (Unknown); Departamento de Salud del Gobierno de Navarra (Unknown)
Responsible Party: Principal Investigator, Jesús Martin, Associate Professor, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HELP-F Study
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Chronic Illness; Caregivers
Keywords: Person-centredness; RCT; Partnership; Health plan; Person-centred care; Person-centered care; Patient-centered care; Home care; In-home care; Home-based care; Community home care; Carers; Family caregivers; Informal caregivers; Care providers
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: Family caregivers of patients with advanced chronic illness who meet the inclusion criteria and provide informed consent will be randomized. Randomization will be conducted at the primary care center level by research nurses, following a computer-generated sequence, with a 1:1 allocation. Centers will be assigned to either the control or intervention group. The control group will receive usual care, while the intervention group will receive a three-month person- and family-centered care intervention, in addition to usual care.
Masking Description: The nature of the intervention means that neither participants nor the health care professionals in the HELP-F intervention can be blinded to allocation in the RCT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants allocated to the control group will not receive any additional intervention. They will continue to receive the standard care provided in primary care for the management of patients with advanced chronic conditions, according to routine clinical practice and regional healthcare guidelines.
- Intervention group (Experimental): The Person-Centred Care intervention will be delivered for 3 months on top of usual care.
  Interventions: Behavioral: Person-centered care intervention

INTERVENTIONS:
Behavioral: Person-centered care intervention — The intervention will be delivered by primary care nurses, in coordination with doctors, social workers, and psychologists from each center. Nurses, previously trained in person-centred care, will collect the family narrative regarding their experiences, needs, goals, and available resources. Based on this, a health plan will be co-created with the family, incorporating short- and long-term objectives, concrete actions, and the supports required. The plan will be reviewed and adapted in monthly follow-up consultations during a three-month period.
  Other Names: PCC
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to learn if a Person-Centred Care (PCC) intervention can improve the caregiving experience and wellbeing of families who provide home care for a loved one with advanced chronic illness. The main questions it aims to answer are:

* Does the PCC intervention improve families' caregiving experience, preparedness for caregiving, and psychological wellbeing?
* Is the PCC intervention feasible and acceptable for implementation in primary care settings?

Researchers will compare families who receive the PCC intervention in addition to usual care to families who receive usual care alone.

Participants will:

* Take part in an initial in-person consultation with a primary care nurse to share their family caregiving experience and co-create a personalized health plan.
* Have monthly follow-up contacts with the same nurse over a 3-month period to update and adapt the plan.
* Receive a copy of the updated plan after each contact to guide caregiving and support decision-making.

DETAILED DESCRIPTION:
BACKGROUND:

More than 4.4 million decedents in Europe experience serious health-related suffering and require palliative care, a number projected to grow globally (Arias-Casais et al., 2019). Although hospital deaths still predominate, deaths at home are steadily increasing (Morris et al., 2015). Importantly, many hospital deaths occur contrary to patients' preferences, as most people would prefer to die at home supported by family (Ali et al., 2019; Gomes et al., 2013; Higginson et al., 2017). In parallel, home-based end-of-life care has expanded in recent years (Arias-Casais et al., 2020; Kjellstadli et al., 2018; Nilsson et al., 2017).

The feasibility of remaining at home near the end of life depends largely on families' capacity to assume caregiving responsibilities (Dowd et al., 2023; Martín-Martín et al., 2022). Family members typically provide most physical and emotional care, symptom management, and service coordination, effectively becoming the backbone of home end-of-life care and delivering ~80% of care for patients with advanced illness at home (Zavagli et al., 2019; Stajduhar, 2013; Martín-Martín et al., 2016; Morris et al., 2015). While home care can foster autonomy, freedom, and meaning (Collier et al., 2015; Akpan-Idiok & Anarado, 2014), it also imposes substantial physical, psychological, and emotional strain on families, who frequently feel unprepared and lack confidence for these roles (Martín-Martín et al., 2016; Mason & Hodgkin, 2019; Soroka et al., 2018).

Health professionals play a crucial role in enabling families to provide sustainable home care in line with preferences for place of care and death (Ewing et al., 2018; Hardy, 2018). Yet family-centred practice often remains aspirational: many services still focus primarily on the patient, and professionals may be unsure how to engage families effectively (Ellington et al., 2018; Lees et al., 2014). Moreover, most research to date has emphasized the individual "primary caregiver," overlooking the broader family unit despite evidence that advanced illness constitutes a family-level crisis requiring collective adjustment during dying and into bereavement (Steele & Davies, 2015; Martín-Martín et al., 2022, 2025; Mehta et al., 2009).

Person-Centred Care (PCC) offers a coherent response. Major organizations-including WHO and the National Academy of Medicine-call for systems that centre the person (and family) rather than the disease (OMS, 2017; Pronovost et al., 2018). Spanish and regional initiatives have similarly promoted person- and family-centred practice and humanization of care (Asociación Profesional de Enfermeras de Ontario, 2015; Departamento de Salud, 2018). PCC, particularly the University of Gothenburg Centre for Person-Centred Care (GPCC) model, organizes care around narratives, shared goals, partnership, and co-creation of a health plan (Ekman et al., 2011; Britten et al., 2020). This approach reframes families as active partners with resources and capabilities, enhancing self-efficacy and participation in decision-making and care planning (Dewing et al., 2021; Barr & Tsai, 2021). Prior frameworks emphasize relational processes and contexts (McCormack & McCance, 2006; Leplège et al., 2007).

Evidence across conditions and settings indicates that PCC can improve self-efficacy, reduce uncertainty and fatigue, shorten hospital stays, lower costs and readmissions, and increase adherence and satisfaction-with signals of cost-effectiveness relative to usual care (Ekman et al., 2012; Dudas et al., 2013; Fors et al., 2017, 2018a; Wallström et al., 2020; Hansson et al., 2016; Sahlen et al., 2016; Brännström & Boman, 2014; Markgren et al., 2019; van Diepen et al., 2020; Leask et al., 2019; Skivington et al., 2024). In advanced illness at home, aligning care with needs and expectations has been associated with improved experiences and outcomes (Ekman et al., 2011; Brännström & Boman, 2014). However, rigorously designed interventions explicitly targeting family units at the end of life remain scarce.

Against this backdrop, the HELP-F project co-designed a PCC intervention tailored to families caring for a loved one with advanced non-oncologic chronic disease at home. A systematic review informed preliminary design, which was then refined via co-design with researchers, primary care professionals, and family caregivers to ensure contextual fit and acceptability (Skivington et al., 2024; Webb et al., 2019).

OBJECTIVES:

General objective: Co-design and pilot a PCC intervention to improve the caregiving experience of families providing home care to a loved one near the end of life, and evaluate feasibility and acceptability of implementation in routine primary care (Asociación Profesional de Enfermeras de Ontario, 2015; Ekman et al., 2011; Britten et al., 2020).

Specific objectives: (1) Co-design the PCC intervention drawing on current evidence and collaboration among researchers, clinicians, and families (Skivington et al., 2024; Webb et al., 2019); (2) Train and assess nurses' PCC competencies as leaders of the intervention (Carvajal-Valcárcel et al., 2024); (3) Explore feasibility and acceptability of implementation from the perspective of intervention nurses to inform a future large-scale RCT (Leask et al., 2019; Skivington et al., 2024).

DESIGN:

Pilot, open-label, multicentre, parallel-group randomized controlled trial with a superiority framework and intention-to-treat comparison (Christensen, 2007; Shah, 2011). Given the risk of contamination, randomization occurs at the cluster (primary care centre) level. The study follows Medical Research Council guidance for development and evaluation of complex interventions; the intervention is considered complex due to multiple interacting components, required skills, heterogeneity of contexts, and the need for flexible tailoring (Skivington et al., 2021, 2024).

SETTING:

Primary Care centres within the public network of the Pamplona health area (Navarra, Spain).

PARTICIPANTS AND RECRUITMENT:

Investigator nurses at participating centres will screen primary care records to identify patient-family units receiving home-based care for advanced chronic disease. Patients will be approached during routine clinic or home visits (or by telephone) to confirm caregiver identification and interest; caregivers will then be contacted, provided study information, and invited to participate. Consent will be obtained prior to any study-related procedures. Cluster allocation (centre = intervention vs control) will be determined before enrolment to guide site-level implementation and minimize cross-arm contamination (Webb et al., 2019; Skivington et al., 2024).

CO-DESIGN OF IMPLEMENTATION A preliminary logic model, derived from the literature and early design work, was iteratively refined through a stakeholder co-design process-including researchers, Navarra primary care professionals, and family caregivers-following best practice to optimize contextual fit, feasibility, and acceptability (Webb et al., 2019; Skivington et al., 2024). Inputs from this process informed practical delivery details (roles, workflows, materials) and anticipated barriers/facilitators within routine primary care.

INTERVENTION Overview and team. The intervention adapts the GPCC PCC model for family units in home end-of-life care (Britten et al., 2020; Ekman et al., 2011). It is led by primary care nurses with support, when indicated, from medicine, social work, and psychology, all operating within a PCC framework (McCormack & McCance, 2006; Leplège et al., 2007).

Preparation and training. Prior to implementation, intervention nurses will complete a 12-hour, in-person training covering PCC principles (GPCC), person-centred communication, motivational/coaching strategies, and the impact of advanced illness on patients, families, and communities. Interactive, practice-oriented methods will be used. During the pilot, monthly micro-refreshers ("training pills") will be emailed to reinforce fidelity. PCC competence will be assessed pre- and post-pilot using the Spanish PCPI-S (Carvajal-Valcárcel et al., 2024).

Core PCC components: (a) Partnership establishment: Nurse and family (and patient, where appropriate) engage as co-experts-family in lived experience; nurse in disciplinary knowledge (Ekman et al., 2011); (b) Narrative elicitation: Using open questions, reflections, and summaries, the nurse facilitates a family narrative about everyday life, caregiving challenges, resources, and priorities (Ekman et al., 2011; Fors et al., 2018b); (c) Co-creation of a personalized health plan: Together they document key topics, short- and long-term goals, concrete actions (what/how/when), internal/external resources, and needed supports (who/how/when). Where relevant, the nurse coordinates with medicine, social work, and psychology to align inputs (Britten et al., 2020; Dewing et al., 2021; Barr & Tsai, 2021).

Contact structure and documentation. An initial in-person consultation initiates the partnership, narrative, and plan; subsequent monthly contacts with the same nurse review and refine the plan, which is shared with families in print or via email to strengthen commitment and continuity (Ekman et al., 2011; Fors et al., 2018b).

FEASIBILITY AND ACCEPTABILITY EVALUATION After the pilot, a structured focus group with intervention nurses-facilitated by the doctoral researcher and a thesis supervisor-will explore implementation feasibility, acceptability, fidelity, contextual barriers/facilitators, strengths, and improvement opportunities, using a predefined guide and qualitative content analysis to inform refinements for a future definitive trial (Leask et al., 2019; Skivington et al., 2024; Elo & Kyngäs, 2008).

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion Criteria for the Person with Advanced Chronic Illness:

   * Diagnosis of an advanced chronic disease, such as chronic heart failure (NYHA functional class IV), renal failure (stages 4-5), chronic obstructive pulmonary disease (COPD) (grades 4-5 on the MRC scale), or liver failure.
   * Not currently receiving care from a specialized palliative care team.
   * Habitual residence in their own home or that of a family member, without requiring permanent hospitalization.
2. Inclusion Criteria for the Family Caregiving Unit:

   * Actively providing care at home to an adult with advanced illness at the time of the study.
   * A minimum of two months must have elapsed since the initiation of family caregiving for the person with advanced chronic illness at home.
   * At least two or more adult family members of the person with advanced illness must participate in the study.
3. Inclusion Criteria for Individual Caregivers

   * Recognized as a caregiver by the person with advanced chronic illness.
   * Aware of the advanced illness diagnosis of the care recipient.
   * Aged 18 years or older.
   * Able to communicate in Spanish.
   * Having the physical and mental capacity to participate in the interview.
   * Willing and able to provide written informed consent to participate in the study.

Exclusion Criteria:

* Life expectancy of less than one year
* Families experiencing an acute crisis situation (e.g., recent bereavement, severe family conflict).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of a PCC intervention on the caregiving experience of family caregivers. | Baseline, 3, 9 months
  The Spanish version of the Scale for End-of-Life Caregiving Appraisal (SEOLCAS) (Hernández-Padilla et al., 2019) will be used. This instrument comprehensively assesses caregivers' experience at the end of life across four domains: physical suffering, caregiving burden, positive appraisal of caregiving, and social support seeking. It comprises 14 items, with total scores categorized as: "low impact" (0-17 points), "moderate impact" (18-40 points), and "high impact" (41-56 points). The Spanish adaptation has demonstrated good internal consistency (α = 0.92).
Evaluate the effect of a PCC intervention on caregivers' preparedness to provide care. | Baseline, 3, 9 months
  The Spanish version of the Caregiver Preparedness Scale (CPS) (Gutierrez-Baena & Romero-Grimaldi, 2021) will be employed. It consists of 8 items evaluating the preparedness of caregivers of vulnerable older adults living at home. Each item is scored on a 5-point Likert scale ranging from 0 (not at all prepared) to 4 (very well prepared), with a total score ranging from 0 to 32; higher scores indicate greater preparedness. The CPS has shown good internal consistency (α = 0.89).

SECONDARY OUTCOMES:
Evaluate the effect of a PCC intervention on caregivers' levels of anxiety and depression. | Baseline, 3, 9 months
  The Spanish version of the Hospital Anxiety and Depression Scale (HADS) (Terol-Cantero et al., 2015) will be used. The instrument consists of 14 items with two subscales: anxiety and depression. Items are rated on a 4-point Likert scale, with higher scores indicating greater severity. Total scores are categorized as: "normal" (0-7), "borderline" (8-10), and "clinical problem" (>11). The Spanish adaptation has been validated in several populations (Costa-Requena et al., 2009; Vallejo et al., 2012), demonstrating good internal consistency (α = 0.83 for anxiety, α = 0.87 for depression) and sensitivity (0.74-0.84) and specificity (0.78-0.80) ranges (Galindo-Vázquez et al., 2015).
Evaluate the effect of a PCC intervention on the perceived burden of family caregivers. | Baseline, 3, 9 months
  The Spanish version of the Zarit Burden Interview (ZBI) (Martín et al., 1996; Odriozola-Gojenola et al., 2008) will be used. This multidimensional questionnaire (physical, emotional-psychological, social, and economic) consists of 22 items rated on a 5-point Likert scale from 0 = "never" to 5 = "almost always." The total score ranges from 22 to 110, classified as: "no burden" (≤46), "mild burden" (47-55), or "severe burden" (≥56). The ZBI has demonstrated high internal consistency (α = 0.92), sensitivity of 98.5%, and specificity of 93.9% (Gort et al., 2005).
Evaluate the effect of a PCC intervention on the quality of life of family caregivers. | Baseline, 3, 9 months
  The Spanish version of the Short Form-12 Health Survey (SF-12) (Alonso et al., 1995; Vilagut et al., 2013) will be used. This instrument comprises 12 items assessing both positive and negative health states across the following domains: physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health. Vilagut et al. (2005) reported adequate consistency, with α > 0.9 for the subscales of physical functioning, role physical, and role emotional, and α = 0.7 for the remaining subscales.

OTHER OUTCOMES:
Evaluate the effect of a PCC intervention on the rate of unplanned hospital admissions. | Baseline, 3, 9 months
  The rate of unplanned hospital admissions related to advanced illness during the intervention and follow-up period will be collected by the assigned nurse from the patient's medical record.
Evaluate the effect of a PCC intervention on the number of unplanned home or primary care visits. | Baseline, 3, 6 months
  The number of unplanned home or primary care visits during the intervention and follow-up period will be extracted from the patient's medical record by the assigned nurse.
Evaluate the effect of a PCC intervention on the place of death of patients with advanced illness. | Baseline, 3, 6 months
  Death due to any cause and the place where it occurred (healthcare institution or home) will be collected by the assigned nurse from the patient's medical record.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Navarra, Facultad de Enfermería, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Webb, R., Rissik, D., Petheram, L., Beh, J. L., & Stafford Smith, M. (2019). Co-designing adaptation decision support: meeting common and differentiated needs. Climatic Change, 153(4), 569-585. https://doi.org/10.1007/s10584-018-2165-7
- [Background] Van Bulck L, Wampers M, Moons P. Research Electronic Data Capture (REDCap): tackling data collection, management, storage, and privacy challenges. Eur J Cardiovasc Nurs. 2022 Jan 11;21(1):85-91. doi: 10.1093/eurjcn/zvab104. PMID 34741600
- [Background] Stajduhar KI. Burdens of family caregiving at the end of life. Clin Invest Med. 2013 Jun 1;36(3):E121-6. doi: 10.25011/cim.v36i3.19722. PMID 23739665
- [Background] Soroka JT, Froggatt K, Morris S. Family Caregivers' Confidence Caring for Relatives in Hospice Care at Home: An Exploratory Qualitative Study. Am J Hosp Palliat Care. 2018 Dec;35(12):1540-1546. doi: 10.1177/1049909118787779. Epub 2018 Jul 11. PMID 29996659
- [Background] Shah PB. Intention-to-treat and per-protocol analysis. CMAJ. 2011 Apr 5;183(6):696; author reply 696. doi: 10.1503/cmaj.111-2033. No abstract available. PMID 21464181
- [Background] Sahlen KG, Boman K, Brannstrom M. A cost-effectiveness study of person-centered integrated heart failure and palliative home care: Based on a randomized controlled trial. Palliat Med. 2016 Mar;30(3):296-302. doi: 10.1177/0269216315618544. Epub 2015 Nov 24. PMID 26603186
- [Background] National Academy of Medicine; The Learning Health System Series; Wang YC, Zenooz A, Sriram RD, Samitt C, Karney M, Johnson W, Goldman J, Gettinger A, Fridsma DB, Bono RC, Palmer S, Johns MME, Pronovost P, editors. Procuring Interoperability: Achieving High-Quality, Connected, and Person-Centered Care. Washington (DC): National Academies Press (US); 2018. Available from http://www.ncbi.nlm.nih.gov/books/NBK594851/ PMID 37733889
- [Background] Organización Mundial de la Salud. (2017). Más sano, más justo, más seguro: la travesía de la salud mundial 2007-2017. Health Journey, 76.
- [Background] Nilsson J, Blomberg C, Holgersson G, Carlsson T, Bergqvist M, Bergstrom S. End-of-life care: Where do cancer patients want to die? A systematic review. Asia Pac J Clin Oncol. 2017 Dec;13(6):356-364. doi: 10.1111/ajco.12678. Epub 2017 Mar 13. PMID 28294576
- [Background] Morris SM, King C, Turner M, Payne S. Family carers providing support to a person dying in the home setting: A narrative literature review. Palliat Med. 2015 Jun;29(6):487-95. doi: 10.1177/0269216314565706. Epub 2015 Jan 29. PMID 25634635
- [Background] Martin-Martin J, Perez-Diez-Del-Corral M, Olano-Lizarraga M, Valencia-Gil S, Saracibar-Razquin MI. Family Narratives About Providing End-of-Life Care at Home. J Fam Nurs. 2022 Feb;28(1):17-30. doi: 10.1177/10748407211025579. Epub 2021 Jun 24. PMID 34165346
- [Background] Markgren R, Brannstrom M, Lundgren C, Boman K. Impacts of person-centred integrated chronic heart failure and palliative home care on pharmacological heart failure treatment: a substudy of a randomised trial. BMJ Support Palliat Care. 2019 Mar;9(1):e10. doi: 10.1136/bmjspcare-2015-000894. Epub 2016 Jan 20. PMID 26792391
- [Background] Leask CF, Sandlund M, Skelton DA, Altenburg TM, Cardon G, Chinapaw MJM, De Bourdeaudhuij I, Verloigne M, Chastin SFM; GrandStand, Safe Step and Teenage Girls on the Move Research Groups. Framework, principles and recommendations for utilising participatory methodologies in the co-creation and evaluation of public health interventions. Res Involv Engagem. 2019 Jan 9;5:2. doi: 10.1186/s40900-018-0136-9. eCollection 2019. PMID 30652027
- [Background] Higginson IJ, Daveson BA, Morrison RS, Yi D, Meier D, Smith M, Ryan K, McQuillan R, Johnston BM, Normand C; BuildCARE. Social and clinical determinants of preferences and their achievement at the end of life: prospective cohort study of older adults receiving palliative care in three countries. BMC Geriatr. 2017 Nov 23;17(1):271. doi: 10.1186/s12877-017-0648-4. PMID 29169346
- [Background] Hansson E, Ekman I, Swedberg K, Wolf A, Dudas K, Ehlers L, Olsson LE. Person-centred care for patients with chronic heart failure - a cost-utility analysis. Eur J Cardiovasc Nurs. 2016 Jun;15(4):276-84. doi: 10.1177/1474515114567035. Epub 2015 Jan 16. PMID 25595358
- [Background] Hardy B. Meeting the needs of carers of people at the end of life. Nurs Stand. 2018 Apr 28;33(1):59-65. doi: 10.7748/ns.2018.e11128. Epub 2018 Mar 27. PMID 29583171
- [Background] García-García, J. A., Reding-Bernal, A., & López-Alvarenga, J. C. (2013). Cálculo del tamaño de la muestra en investigación en educación médica. Investigación En Educación Médica, 2(8), 217-224. https://doi.org/10.1016/S2007-5057(13)72715-7
- [Background] Fors A, Blanck E, Ali L, Ekberg-Jansson A, Fu M, Lindstrom Kjellberg I, Makitalo A, Swedberg K, Taft C, Ekman I. Effects of a person-centred telephone-support in patients with chronic obstructive pulmonary disease and/or chronic heart failure - A randomized controlled trial. PLoS One. 2018 Aug 31;13(8):e0203031. doi: 10.1371/journal.pone.0203031. eCollection 2018. PMID 30169539
- [Background] Ewing G, Austin L, Jones D, Grande G. Who cares for the carers at hospital discharge at the end of life? A qualitative study of current practice in discharge planning and the potential value of using The Carer Support Needs Assessment Tool (CSNAT) Approach. Palliat Med. 2018 May;32(5):939-949. doi: 10.1177/0269216318756259. Epub 2018 Feb 28. PMID 29490198
- [Background] Ekman I, Swedberg K, Taft C, Lindseth A, Norberg A, Brink E, Carlsson J, Dahlin-Ivanoff S, Johansson IL, Kjellgren K, Liden E, Ohlen J, Olsson LE, Rosen H, Rydmark M, Sunnerhagen KS. Person-centered care--ready for prime time. Eur J Cardiovasc Nurs. 2011 Dec;10(4):248-51. doi: 10.1016/j.ejcnurse.2011.06.008. Epub 2011 Jul 20. PMID 21764386
- [Background] Departamento de Salud. (2018). Estrategia de humanización del Sistema Sanitario Público de Navarra. . Departamento de Salud. Gobierno de Navarra.
- [Background] Christensen E. Methodology of superiority vs. equivalence trials and non-inferiority trials. J Hepatol. 2007 May;46(5):947-54. doi: 10.1016/j.jhep.2007.02.015. Epub 2007 Mar 9. PMID 17412447
- [Background] Carvajal-Valcarcel A, Benitez E, Lizarbe-Chocarro M, Galan-Espinilla MJ, Vazquez-Calatayud M, Errasti-Ibarrondo B, Choperena A, McCormack B, Tyagi V, La Rosa-Salas V. Translation, Cultural Adaptation, and Validation of the Spanish Version of the Person-Centred Practice Inventory-Staff (PCPI-S). Healthcare (Basel). 2024 Dec 9;12(23):2485. doi: 10.3390/healthcare12232485. PMID 39685107
- [Background] Britten N, Ekman I, Naldemirci O, Javinger M, Hedman H, Wolf A. Learning from Gothenburg model of person centred healthcare. BMJ. 2020 Sep 1;370:m2738. doi: 10.1136/bmj.m2738. No abstract available. PMID 32873594
- [Background] Asociación Profesional de Enfermeras de Ontario. (2015). Cuidados centrados en la persona y familia. Investén ISCIII.
- [Background] Arias-Casais N, Lopez-Fidalgo J, Garralda E, Pons JJ, Rhee JY, Lukas R, de Lima L, Centeno C. Trends analysis of specialized palliative care services in 51 countries of the WHO European region in the last 14 years. Palliat Med. 2020 Sep;34(8):1044-1056. doi: 10.1177/0269216320931341. Epub 2020 Jun 10. PMID 32519584
- [Background] Arias-Casais, N., Garralda, E., Rhee, J. Y., Lima, L., Pons-Izquierdo, J. J., Clark, D., Hasselaar, J., Ling, J., Mosoiu, D., & Centeno, C. (2019). EAPC Atlas of Palliative Care in Europe 2019. EAPC Press.
- [Background] Ali M, Capel M, Jones G, Gazi T. The importance of identifying preferred place of death. BMJ Support Palliat Care. 2019 Mar;9(1):84-91. doi: 10.1136/bmjspcare-2015-000878. Epub 2015 Sep 25. PMID 26408428